CLINICAL TRIAL: NCT01822106
Title: Randomized, Double Blind, Placebo Control Trial to Evaluate the Efficacy of Wu-Chu-Yu Tang on Gastroesophageal Reflux Disease (GERD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH102-REC2-011
Record Dates: First submitted 2013-03-24; First posted 2013-04-02 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omeprazole (Active Comparator): Omeprazole at a rate of 20mg once per day
  Interventions: Other: Placebo
- Wu-Chu-Yu Tang (Experimental): Wu-Chu-Yu Tang at a rate of 3.0 g three times per day
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo

SUMMARY:
GERD is due to gastric content reflux to esophagus cause symptom and complication including intra-esophagus such as reflux esophagitis, and extra-esophagus such as cough etc. Because the changes of dietary habit, and improvement of examination skill and data analysis, the prevalence of GERD increased 2.5 multiple from 1995 to 2002, and suggesting the prevalence is 25% in Taiwan community.

Although proton pump inhibitor (PPI) can inhibit gastric acid secretion, relief symptom and enhancing repair of esophageal damage, therefore, PPI is a main drug for the treatment of GRED, but because of PPI has disadvantage of poor compliance, and slow gastric empty time and hypersensitivity, and about 40-50% of GERD patients is inefficacy. In addition, PPI produces bone fracture, community pneumonia and diarrhea in patient with long-term use.

Wu-Chu-Yu tang consists of Evodia fargesii Dode (Evodia Fruit), Panax ginseng C. (Ginseng), Ziziphus jujube Mill (Chinses Date), Zingiber officinale Rosee (Fresh Ginger). According to "I-Fang-Chi-Chieh" and "Shanghonzobinglun" recordings that Wu-Chu-Yu tang can treat vomiting, and also can relax gastric tonicity and can enhance peristalsis of stomach.

Therefore, the purpose of the present study was to investigate the efficacy of Wu-Chu-Yu tang on GRED, and this effect of Wu-Chu-Yu tang compared to PPI Omeprazole.

ELIGIBILITY:
Inclusion Criteria:

1. Gender:Male or female.
2. Age: from 20 y/o to 75 y/o.
3. The diagnosis is Gastroesophageal Reflux Disease.
4. With the symptoms of heartburn or acid regurgitation.
5. After explaining thoroughly the whole research purpose or process, the clients are willing to sign the agreement.

Exclusion Criteria:

1. Exclude peptic ulcer, gall bladder stone (including intraheptaic and common hepatical duct) and major diseased of cancer.
2. Barrett's esophagus or esophagus stricture.
3. The operation history of esophagus or gastroduodenoal regions.
4. Tarry stool suspected GI tract bleeding.
5. With the history of alcohol or drug abuse.
6. The clients with the history of study drug allergy.
7. The clients with psychologic cannot cooperate with each other.
8. The pregnant woman or the lactating women.
9. Abnormal liver function such as GOT, GPT elevated over double the normal range.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
RDQ Questionnaire | Chang from baseline RDQ score at week 4 (28 ± 5 days)

SECONDARY OUTCOMES:
GerD Questionnaire | Chang from baseline GerD score at week 4 (28 ± 5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Hsueh Chou Lai, MD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan